CLINICAL TRIAL: NCT05981417
Title: Effect of a Physiotherapy Intervention Based on Therapeutic Exercise on the Psychological Well-being of Women Victims of Gender Violence.
Brief Title: Therapeutic Exercise on the Psychological Well-being of Women Victims of Gender Violence.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Collaborators: Centro de Información Municipal á Muller de Poio (Unknown); Centro de Información Municipal á Muller de Pontevedra (Unknown)
Responsible Party: Principal Investigator, Lorenzo Antonio Justo Cousino, PhD, Physical Therapist, PhD., University of Vigo
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UVigo
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Anxiety Disorders; Depressive Symptoms; Gender-based Violence
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised exercise (Experimental): Exercise sessions will beguided by a physiotherapist.
  Interventions: Other: Therapeutic exercise
- Home exercise (Active Comparator): Exercise sessions will be perfomed at home.
  Interventions: Other: Therapeutic exercise

INTERVENTIONS:
Other: Therapeutic exercise — Therapeutic exercise sessions will be guided by a physiotherapist.
  Arms: Supervised exercise
Other: Therapeutic exercise — Therapeutic exercise sessions will be performed at home.
  Arms: Home exercise

SUMMARY:
The scientific literature shows that women subjected to gender violence suffer a deterioration in mental health (anxiety, stress and depression). In particular, a recent study carried out in Galicia found a high incidence of post-traumatic stress, depression and low self-esteem in women victims of gender violence.

The efficacy of therapeutic exercise in depression and anxiety has been widely demonstrated, as has the link between gender violence and deterioration of mental health, with a high incidence of post-traumatic stress. However, research on the effect of therapeutic exercise in battered women is very limited.

For this reason, the aim of the present project is to evaluate the effect of a therapeutic exercise program on mental health in women who have suffered gender violence.

ELIGIBILITY:
Inclusion Criteria:

* Women of legal age with a history of gender-based violence who come to the women's center or are included in the women's center's programs.

Exclusion Criteria:

* Consumption of alcohol or other drugs.
* Musculoskeletal disorders, recent surgery, as well as any physical problem that prevents exercise.
* Any medical contraindication to exercise.
* Pregnancy.
* Having any affirmative answer in the PARQ questionnaire (Physical Activity Readiness Questionnaire).
* Participants who do not have the capacity to consent to participate will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Psychological well-being assessed by Ryff psychological well-being scale. | 8 weeks
  This self-report instrument consist of a series of statements reflecting the six areas of psychological well-being: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. Respondents rate statements on a scale of 1 to 6, with 1 indicating strong disagreement and 6 indicating strong agreement.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - University of Vigo, Pontevedra
  - Lorenzo Justo Cousiño, Pontevedra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dragesund T, Raheim M. Norwegian psychomotor physiotherapy and patients with chronic pain: patients' perspective on body awareness. Physiother Theory Pract. 2008 Jul-Aug;24(4):243-54. doi: 10.1080/09593980701738400. PMID 18574750
- [Background] Friis S, Skatteboe UB, Hope MK, Vaglum P. Body awareness group therapy for patients with personality disorders. 2. Evaluation of the Body Awareness Rating Scale. Psychother Psychosom. 1989;51(1):18-24. doi: 10.1159/000288129. PMID 2602528
- [Background] Strohle A. Sports psychiatry: mental health and mental disorders in athletes and exercise treatment of mental disorders. Eur Arch Psychiatry Clin Neurosci. 2019 Aug;269(5):485-498. doi: 10.1007/s00406-018-0891-5. Epub 2018 Mar 21. PMID 29564546
- [Background] Smith PJ, Merwin RM. The Role of Exercise in Management of Mental Health Disorders: An Integrative Review. Annu Rev Med. 2021 Jan 27;72:45-62. doi: 10.1146/annurev-med-060619-022943. Epub 2020 Nov 30. PMID 33256493
- [Background] Carek PJ, Laibstain SE, Carek SM. Exercise for the treatment of depression and anxiety. Int J Psychiatry Med. 2011;41(1):15-28. doi: 10.2190/PM.41.1.c. PMID 21495519
- [Background] Ross RE, VanDerwerker CJ, Saladin ME, Gregory CM. The role of exercise in the treatment of depression: biological underpinnings and clinical outcomes. Mol Psychiatry. 2023 Jan;28(1):298-328. doi: 10.1038/s41380-022-01819-w. Epub 2022 Oct 17. PMID 36253441
- [Background] Schuch FB, Vancampfort D. Physical activity, exercise, and mental disorders: it is time to move on. Trends Psychiatry Psychother. 2021 Jul-Sep;43(3):177-184. doi: 10.47626/2237-6089-2021-0237. Epub 2021 Apr 21. PMID 33890431
- [Background] Herring MP, Jacob ML, Suveg C, Dishman RK, O'Connor PJ. Feasibility of exercise training for the short-term treatment of generalized anxiety disorder: a randomized controlled trial. Psychother Psychosom. 2012;81(1):21-8. doi: 10.1159/000327898. Epub 2011 Nov 22. PMID 22116310
- [Background] Jonker IE, Lako DAM, Beijersbergen MD, Sijbrandij M, van Hemert AM, Wolf JRLM. Factors Related To Depression and Post-Traumatic Stress Disorder in Shelter-Based Abused Women. Violence Against Women. 2019 Mar;25(4):401-420. doi: 10.1177/1077801218790700. Epub 2018 Aug 20. PMID 30124130
- [Background] Mondolfi Miguel ML, Rosa Pino-Juste M. Psycho-social profile of battered women in Galicia, Spain: Distress as a result of intimate partner violence and child abuse. Health Care Women Int. 2019 Nov;40(11):1229-1248. doi: 10.1080/07399332.2019.1571061. Epub 2019 Feb 12. PMID 30753120
- [Background] Dunn AL, Trivedi MH, Kampert JB, Clark CG, Chambliss HO. Exercise treatment for depression: efficacy and dose response. Am J Prev Med. 2005 Jan;28(1):1-8. doi: 10.1016/j.amepre.2004.09.003. PMID 15626549
- [Background] Gordon BR, McDowell CP, Lyons M, Herring MP. Resistance exercise training for anxiety and worry symptoms among young adults: a randomized controlled trial. Sci Rep. 2020 Oct 16;10(1):17548. doi: 10.1038/s41598-020-74608-6. PMID 33067493